CLINICAL TRIAL: NCT02424994
Title: Morbidity and Mortality in Patients Diagnosed With Hypertrophic Cardiomyopathy: a CALIBER Study
Brief Title: Morbidity and Mortality in Patients With Hypertrophic Cardiomyopathy: a CALIBER Study
Acronym: HCM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Inherited Cardiac Diseases Unit, The Heart Hospital, London (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13_096R
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Morbidity; Mortality; Health care utilization; Cohort; Epidemiology; Cardiovascular diseases
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Patient Acceptance of Health Care; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
The aim of this project is to study the association of a number of demographic and cardiovascular risk factors with death, health care utilisation and systemic embolisation by examining the clinical evolution of hypertrophic cardiomyopathy in a large, community based cohort identified from linked electronic health records.

DETAILED DESCRIPTION:
Most data on hypertrophic cardiomyopathy related morbidity and mortality are derived primarily from longitudinal, observational studies based at tertiary cardiac centres. It is unclear what the main causes of morbidity and death are in the general hypertropic cardiomyopathy population (outside tertiary referral centres) and it is likely that many patients have a benign clinical course and die from non-cardiac causes.

Linkage of the Clinical Practice Research Datalink (CPRD) to the Myocardial Ischaemia National Audit Project (MINAP), Hospital Episode Statistics (HES) and Office of National Statistics (ONS), offers the opportunities to study the natural history of hypertrophic cardiomyopathy, from the time of diagnosis to the end of life, health care utilisation and to investigate the association between clinical characteristics and common clinical fatal and non-fatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* One year or more of follow-up in the practice prior to study entry
* 18 years or older

Exclusion Criteria:

• Unknown sex and age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients registered in Clinical Practice Research Datalink (CPRD) practices
Sampling Method: Non-Probability Sample
Enrollment: 12464 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Rate ratios for the associations between hypertrophic cardiomyopathy and angina | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and unstable angina | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and myocardial infarction | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and coronary heart disease not otherwise specified | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and cardiac arrest | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and ventricular arrhythmia | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and atrial fibrillation | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and heart failure | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and transient ischemic attack | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and stroke | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and peripheral arterial disease | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and abdominal aortic aneurysm | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and systemic thromboembolism | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)

SECONDARY OUTCOMES:
Rate ratios for the associations between hypertrophic cardiomyopathy and cancer | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and chronic obstructive pulmonary disease | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)
Rate ratios for the associations between hypertrophic cardiomyopathy and liver-related | Followed for the duration of general practice registration between date of eligibility and date of administrative censoring, outcome occurrence or death (expected median of 4 years)

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Farr Institute of Health Informatics Research, London, United Kingdom